CLINICAL TRIAL: NCT01906034
Title: Effects of a Fall Preventive Exercise Program on Intrinsic Fall Risk Factors in Healthy Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Potsdam (Other)
Collaborators: Swiss Council for Accident Prevention (Unknown); Prof. Dr. Reto W. Kressig and Dr. Yves Gschwind, University Center for Medicine of Aging Basel (UAB), Felix Platter-Hospital, Basel, Switzerland (Unknown)
Responsible Party: Principal Investigator, Urs Granacher, PhD, University of Potsdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFU-2.104
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Fall Risk Factors; Fall Prevention
MeSH Terms: interventions — Exercise; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise with supervision (Experimental): The expert panel selected balance and strength / power exercises which can be performed with one's own bodyweight or with the help of small, low-cost exercise equipment (i.e., small weights, resistance bands, unstable surfaces). In this study, intensity during training will be regulated using the Borg Rating of Perceived Exertion scale (i.e., 6-20 points, maximal exertion at 20 points). According to the individual fitness level, exercises should be performed with a perceived exertion between 12 and 16 points (somewhat hard - hard) during balance and strength / power training. Exercise intensity will be progressed individually using the Borg Rating of Perceived Exertion scale and varying the balance and strength / power exercises in order to sufficiently stimulate the neuromuscular system. Strength / power exercises will be progressed from single to multiple joint, isometric to dynamic muscle contraction, short to long lever arm and slow to fast exercises.
  Interventions: Behavioral: Exercise with supervision
- Home-based without supervision (Experimental): The expert panel selected balance and strength / power exercises which can be performed with one's own bodyweight or with the help of small, low-cost exercise equipment (i.e., small weights, resistance bands, unstable surfaces). In this study, intensity during training will be regulated using the Borg Rating of Perceived Exertion scale (i.e., 6-20 points, maximal exertion at 20 points). According to the individual fitness level, exercises should be performed with a perceived exertion between 12 and 16 points (somewhat hard - hard) during balance and strength / power training. Exercise intensity will be progressed individually using the Borg Rating of Perceived Exertion scale and varying the balance and strength / power exercises in order to sufficiently stimulate the neuromuscular system. Strength / power exercises will be progressed from single to multiple joint, isometric to dynamic muscle contraction, short to long lever arm and slow to fast exercises.
  Interventions: Behavioral: Home-based without supervision
- control group (No Intervention): The control group is a traditional waiting group and will receive a supervised training program after the completion of this study

INTERVENTIONS:
Behavioral: Exercise with supervision
  Arms: Exercise with supervision
Behavioral: Home-based without supervision
  Arms: Home-based without supervision

SUMMARY:
Background With increasing age neuromuscular deficits (e.g., sarcopenia) may result in impaired physical performance and an increased risk for falls. Prominent intrinsic fall-risk factors are age-related decreases in balance and strength / power performance as well as cognitive decline. Additional studies are needed to develop specifically tailored exercise programs for older adults that can easily be implemented into clinical practice. Thus, the objective of the present trial is to assess the effects of a fall prevention program that was developed by an interdisciplinary expert panel on measures of balance, strength / power, body composition, cognition, psychosocial well-being, and falls self-efficacy in healthy older adults. Additionally, the time-related effects of detraining are tested.

Methods/Design Healthy old people (N = 66) between the age of 65 to 80 years will participate in this trial. The testing protocol comprises tests for the assessment of static / dynamic steady-state balance (i.e., Sharpened Romberg Test, instrumented gait analysis), proactive balance (i.e., Functional Reach Test; Timed Up and Go Test), reactive balance (i.e., perturbation test during bipedal stance; Push and Release Test), strength (i.e., hand grip strength test; Chair Stand Test), and power (i.e., Stair Climb Power Test). Further, body composition will be analysed using a bioelectrical impedance analysis system. In addition, questionnaires for the assessment of psychosocial (i.e., World Health Organisation Quality of Life Assessment-Bref), cognitive (i.e., Mini Mental State Examination), and fall risk determinants (i.e., Fall Efficacy Scale - International) will be included in the study protocol. Participants will be randomized into two intervention groups or the control / waiting group. After baseline measures, participants in the intervention groups will conduct a 12-week balance and strength / power exercise intervention 3 times per week, with each training session lasting 30 min (without warm-up and cool-down). One intervention group will complete a supervised training program (2x supervised training per week / 1x home training per week), while the other intervention group will complete a training after the same protocol that is home-based (3x home training per week) and controlled by phone calls every two weeks. Post-tests will be conducted right after the intervention period. Additionally, detraining effects will be measured 12 weeks after program cessation. The control group / waiting group will not participate in any specific intervention during the experimental period, but will receive the extensive supervised program after the experimental period.

Discussion It is expected that particularly the supervised combination of balance and strength / power training will improve performance in variables of balance, strength / power, body composition, cognitive function, psychosocial well-being, and falls self-efficacy of older adults. In addition, information regarding fall risk assessment, detraining effects, and supervision of training will be provided. Further, training-induced health-relevant changes, such as improved performance in activities of daily living, cognitive function, and quality of life, as well as a reduced risk for falls may help to lower costs in the health care system. Finally, practitioners, therapists, and instructors will be provided with a scientifically evaluated, feasible, safe, and easy-to-administer exercise program for fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years old
* must be able to accomplish the tests and the training
* must be able to walk independently

Exclusion Criteria:

* neurological diseases: Alzheimer´s disease, Multiple Sclerosis, Parkinson etc.
* cardiovascular diseases: coronary heart disease, cardiac arrhythmias etc.
* artificial knee- hip-joint in the last six months
* regular participation in strength and/or balance training programs
* acute injuries impairing the tests
* disturbances of balance

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Balance Performance, Strength / Power Performance | pre, post (12 weeks) and follow-up (24 weeks)

SECONDARY OUTCOMES:
cognitive status, psychosocial health, falls efficacy | pre, post (12 weeks) and follow-up (24 weeks)

OTHER OUTCOMES:
body composition | pre, post (12 weeks) and follow-up (24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Urs Granacher, PhD, Principal Investigator — University of Potsdam, Department of Training and Movement Science; Andre Lacroix, Master, Study Chair — University of Potsdam, Department of Training and Movement Science
Locations (1):
- University of Potsdam, Department of Training and Movement Sciences, Potsdam, Germany

REFERENCES:
- [Background] Granacher U, Muehlbauer T, Gruber M. A qualitative review of balance and strength performance in healthy older adults: impact for testing and training. J Aging Res. 2012;2012:708905. doi: 10.1155/2012/708905. Epub 2012 Jan 23. PMID 22315687
- [Background] Granacher U, Muehlbauer T, Zahner L, Gollhofer A, Kressig RW. Comparison of traditional and recent approaches in the promotion of balance and strength in older adults. Sports Med. 2011 May 1;41(5):377-400. doi: 10.2165/11539920-000000000-00000. PMID 21510715
- [Background] Granacher U, Gruber M, Gollhofer A. Resistance training and neuromuscular performance in seniors. Int J Sports Med. 2009 Sep;30(9):652-7. doi: 10.1055/s-0029-1224178. Epub 2009 Jun 30. PMID 19569007
- [Background] Granacher U, Gollhofer A, Strass D. Training induced adaptations in characteristics of postural reflexes in elderly men. Gait Posture. 2006 Dec;24(4):459-66. doi: 10.1016/j.gaitpost.2005.12.007. Epub 2006 Feb 2. PMID 16472525
- [Background] Granacher U, Gollhofer A, Hortobagyi T, Kressig RW, Muehlbauer T. The importance of trunk muscle strength for balance, functional performance, and fall prevention in seniors: a systematic review. Sports Med. 2013 Jul;43(7):627-41. doi: 10.1007/s40279-013-0041-1. PMID 23568373
- [Background] Beijersbergen CM, Granacher U, Vandervoort AA, DeVita P, Hortobagyi T. The biomechanical mechanism of how strength and power training improves walking speed in old adults remains unknown. Ageing Res Rev. 2013 Mar;12(2):618-27. doi: 10.1016/j.arr.2013.03.001. Epub 2013 Mar 15. PMID 23501431
- [Background] Granacher U, Lacroix A, Muehlbauer T, Roettger K, Gollhofer A. Effects of core instability strength training on trunk muscle strength, spinal mobility, dynamic balance and functional mobility in older adults. Gerontology. 2013;59(2):105-13. doi: 10.1159/000343152. Epub 2012 Oct 24. PMID 23108436
- [Background] Muehlbauer T, Besemer C, Wehrle A, Gollhofer A, Granacher U. Relationship between strength, power and balance performance in seniors. Gerontology. 2012;58(6):504-12. doi: 10.1159/000341614. Epub 2012 Aug 24. PMID 22922168
- [Background] Muehlbauer T, Roth R, Bopp M, Granacher U. An exercise sequence for progression in balance training. J Strength Cond Res. 2012 Feb;26(2):568-74. doi: 10.1519/JSC.0b013e318225f3c4. PMID 22067238
- [Background] Granacher U, Bridenbaugh SA, Muehlbauer T, Wehrle A, Kressig RW. Age-related effects on postural control under multi-task conditions. Gerontology. 2011;57(3):247-55. doi: 10.1159/000322196. Epub 2010 Oct 27. PMID 20980734
- [Background] Granacher U, Muehlbauer T, Bridenbaugh S, Bleiker E, Wehrle A, Kressig RW. Balance training and multi-task performance in seniors. Int J Sports Med. 2010 May;31(5):353-8. doi: 10.1055/s-0030-1248322. Epub 2010 Feb 23. PMID 20180173
- [Background] Granacher U, Gruber M, Gollhofer A. Force production capacity and functional reflex activity in young and elderly men. Aging Clin Exp Res. 2010 Oct-Dec;22(5-6):374-82. doi: 10.1007/BF03337733. Epub 2009 Nov 27. PMID 19966537
- [Result] Lacroix A, Kressig RW, Muehlbauer T, Gschwind YJ, Pfenninger B, Bruegger O, Granacher U. Effects of a Supervised versus an Unsupervised Combined Balance and Strength Training Program on Balance and Muscle Power in Healthy Older Adults: A Randomized Controlled Trial. Gerontology. 2016;62(3):275-88. doi: 10.1159/000442087. Epub 2015 Dec 9. PMID 26645282
- [Derived] Gschwind YJ, Kressig RW, Lacroix A, Muehlbauer T, Pfenninger B, Granacher U. A best practice fall prevention exercise program to improve balance, strength / power, and psychosocial health in older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2013 Oct 9;13:105. doi: 10.1186/1471-2318-13-105. PMID 24106864